CLINICAL TRIAL: NCT03947255
Title: A Phase 2, Multicenter, Single-arm Study of Retreatment With Brentuximab Vedotin in Subjects With Relapsed or Refractory Classic Hodgkin Lymphoma (cHL) or CD30-expressing Peripheral T Cell Lymphoma (PTCL)
Brief Title: A Study of Retreatment With Brentuximab Vedotin in Subjects With Classic Hodgkin Lymphoma or CD30-expressing Peripheral T Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped early due to low patient accrual.
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-028
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Hodgkin Lymphoma; Peripheral T Cell Lymphoma; Anaplastic Large Cell Lymphoma
Keywords: CD30-expression; sALCL; PTCL; cHL; Seattle Genetics
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, T-Cell, Peripheral; Lymphoma, Large-Cell, Anaplastic | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brentuximab vedotin (Experimental)
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg given intravenously (IV)
  Other Names: ADCETRIS; SGN-35

SUMMARY:
This study will look at whether brentuximab vedotin works and is safe in the re-treatment setting. To be in this study, patients must have already received brentuximab vedotin as treatment and have cancer that progressed (got worse) after stopping treatment.

DETAILED DESCRIPTION:
This is a study to determine the safety and efficacy of brentuximab vedotin in subjects with classic Hodgkin lymphoma (cHL) and systemic anaplastic large cell lymphoma (sALCL) or other CD30-expressing peripheral T cell lymphoma (PTCL) who experienced complete response (CR) or partial response (PR) with a brentuximab vedotin-containing regimen and subsequently experienced disease progression or relapse.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cHL, sALCL, or other CD30-expressing PTCL
* Previously treated with brentuximab vedotin containing regimen, with evidence of objective response, and subsequent disease progression or relapse after discontinuing treatment
* Documentation of disease relapse or progression ≥6 months after the last dose of brentuximab vedotin
* Fluorodeoxyglucose positron emission tomography- (FDG-PET) avid and bidimensional measurable disease of at least 1.5 cm in longest axis as documented by radiographic technique
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2
* Must not be pregnant and, if of childbearing or fathering potential, must agree to use 2 effective contraception methods during study and for 6 months following last dose of study drug

Exclusion Criteria:

* Previously discontinued brentuximab vedotin due to any Grade 3 or higher toxicity
* Existing Grade 2 or higher peripheral neuropathy
* Previously refractory to treatment with brentuximab vedotin
* History of a cerebral vascular event, unstable angina, or myocardial infarction within 6 months prior to first dose
* History of another malignancy within 3 years before first dose of study drug or any evidence of residual disease from previously diagnosed malignancy
* Acute or chronic graft-versus-host-disease (GvHD) or receiving immunosuppressive therapy as treatment for or prophylaxis agent against GvHD
* Active cerebral/meningeal disease
* History of progressive multifocal leukoencephalopathy (PML)
* Active uncontrolled Grade 3 (per NCI CTCAE v5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to first dose of study drug
* Chemotherapy, radiotherapy, biologics, and/or other antitumor treatment with immunotherapy that is not completed 4 weeks prior to first dose of study drug, unless underlying disease has progressed on treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Lai, MD, Study Director — Seagen Inc.
Locations (19):
- United States (19):
  - Pacific Cancer Medical Center, Anaheim, California
  - SCL Health Good Samaritan Medical Center Cancer Centers of Colorado, Lafayette, Colorado
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - Northwest Oncology and Hematology/AMITA, Elk Grove Village, Illinois
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Saint Louis University, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Summit Medical Group, Florham Park, New Jersey
  - Medical University of South Carolina/Hollings Cancer Center, Charleston, South Carolina
  - Texas Oncology - Fort Worth, Dallas, Texas
  - Texas Oncology - Fort Worth 12th Avenue, Fort Worth, Texas
  - The Center for Cancer and Blood Disorders: Fortworth, Fort Worth, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Classic Hodgkin Lymphoma: Participants with classic Hodgkin lymphoma
- PTCL: Participants with peripheral T cell lymphoma
Period: Overall Study
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Study Closure by Sponsor | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set includes participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Classic Hodgkin Lymphoma | PTCL | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 0 | 3 | 3
Age, Continuous [Median (Full Range); unit: Years] | 31 [28 to 55] | 63 [35 to 77] | 50 [28 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — Measure Description: 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead
  Participants
    Grade 0 | 3 | 2 | 5
    Grade 1 | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per BICR According to Modified Lugano Response Criteria
Description: Objective Response Rate (ORR) is defined as the percentage of participants with complete response (CR) or partial response (PR) according to the modified Lugano Criteria for Response Assessment (Cheson 2014) based on BICR
Time Frame: Up to 18.3 months
Population: The full analysis set includes participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 5 | 6
percentage of participants | 40.0 [5.3 to 85.3] | 83.3 [35.9 to 99.6]

2. Primary Outcome: Number of Participants With Adverse Events
Description: An AE is any untoward medical occurrence in a patient or clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Treatment emergent AEs (TEAEs) are defined as events that are new or worsened on or after receiving the first dose of study treatment and up through 30 days after the last dose of study treatment.
Time Frame: Up to 36 months
Population: The full analysis set includes participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 5 | 6
Participants
  Any TEAE | 5 | 6
  Treatment-related TEAE | 4 | 5
  Any Treatment-Emergent SAE | 0 | 2
  Discontinuation of treatment due to TEAE | 1 | 3
  Discontinuation of treatment due to treatment-related TEAE | 1 | 3
  TEAE leading to death | 0 | 0

3. Secondary Outcome: Duration of Response (DOR) Per BICR According to Modified Lugano Response Criteria
Description: Duration of response is defined as the time from start of the first documentation of objective tumor response (CR or PR), according to the Modified Lugano Criteria for Response Assessment (Cheson 2007), to the first documentation of objective tumor progression or to death due to any cause, whichever comes first.
Time Frame: Up to 17.1 months
Population: The full analysis set includes participants who received at least one dose of study treatment. This is a subset analysis of participants with complete response or partial response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 2 | 5
months | NA [NA to NA] — Not enough events to calculate Median or Lower and Upper Limits. | NA [2.9 to NA] — Not enough events to calculate Median or Upper Limit.

4. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory data was summarized by the worst post-baseline grade, by NCI CTCAE v5.0 or higher for each parameter.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 5 | 6
Participants
  Hemoglobin Low, Grade 1-2 | 3 | 2
  Hemoglobin Low, Grade 3 | 0 | 0
  Hemoglobin Low, Grade 4 | 0 | 0
  Leukocytes Low, Grade 1-2 | 1 | 2
  Leukocytes Low, Grade 3 | 0 | 0
  Leukocytes Low, Grade 4 | 0 | 0
  Lymphocytes Low, Grade 1-2 | 1 | 1
  Lymphocytes Low, Grade 3 | 0 | 1
  Lymphocytes Low, Grade 4 | 0 | 0
  Neutrophils Low, Grade 1-2 | 0 | 2
  Neutrophils Low, Grade 3 | 0 | 1
  Neutrophils Low, Grade 4 | 0 | 0
  Platelets Low, Grade 1-2 | 1 | 2
  Platelets Low, Grade 3 | 0 | 0
  Platelets Low, Grade 4 | 0 | 0
  Alanine Aminotransferase High, Grade 1-2 | 1 | 0
  Alanine Aminotransferase High, Grade 3 | 0 | 0
  Alanine Aminotransferase High, Grade 4 | 0 | 0
  Albumin Low, Grade 1-2 | 0 | 3
  Albumin Low, Grade 3 | 0 | 0
  Albumin Low, Grade 4 | 0 | 0
  Alkaline Phosphatase High, Grade 1-2 | 1 | 3
  Alkaline Phosphatase High, Grade 3 | 0 | 0
  Alkaline Phosphatase High, Grade 4 | 0 | 0
  Aspartate Aminotransferase High, Grade 1-2 | 3 | 2
  Aspartate Aminotransferase High, Grade 3 | 0 | 0
  Aspartate Aminotransferase High, Grade 4 | 0 | 0
  Bilirubin High, Grade 1-2 | 0 | 1
  Bilirubin High, Grade 3 | 0 | 0
  Bilirubin High, Grade 4 | 0 | 0
  Calcium Corrected for Albumin Low, Grade 1-2 | 0 | 1
  Calcium Corrected for Albumin Low, Grade 3 | 0 | 0
  Calcium Corrected for Albumin Low, Grade 4 | 0 | 0
  Creatinine High, Grade 1-2 | 1 | 1
  Creatinine High, Grade 3 | 0 | 1
  Creatinine High, Grade 4 | 0 | 0
  Lactate Dehydrogenase High, Grade 1-2 | 3 | 4
  Lactate Dehydrogenase High, Grade 3 | 0 | 0
  Lactate Dehydrogenase High, Grade 4 | 0 | 0
  Potassium Low, Grade 1-2 | 1 | 2
  Potassium Low, Grade 3 | 0 | 1
  Potassium Low, Grade 4 | 0 | 0
  Sodium High, Grade 1-2 | 0 | 1
  Sodium High, Grade 3 | 0 | 0
  Sodium High, Grade 4 | 0 | 0
  Sodium Low, Grade 1-2 | 3 | 1
  Sodium Low, Grade 3 | 0 | 0
  Sodium Low, Grade 4 | 0 | 0

5. Secondary Outcome: Progression-free Survival (PFS) Per BICR According to Modified Lugano Response Criteria
Description: PFS is defined as the time from start of study treatment to first documentation of objective tumor progression according to the Modified Lugano Criteria for Response Assessment (Cheson 2007) or to death due to any cause, whichever comes first.
Time Frame: up to 18.3 months
Population: The full analysis set includes participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 5 | 6
Months | NA [1.3 to NA] — Not enough events to calculate Median or Upper Limit. | NA [1.1 to NA] — Not enough events to calculate Median or Upper Limit.

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of enrollment to date of death due to any cause.
Time Frame: Up to 35.8 months
Population: The full analysis set includes participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 5 | 6
Months | NA [NA to NA] — Not enough events to calculate Median or Lower and Upper Limits. | NA [1.1 to NA] — Not enough events to calculate Median or Upper Limit.

7. Secondary Outcome: Rate of Complete Response (CR) Per BICR According to Modified Lugano Response Criteria
Description: CR rate is defined as the percentage of participants with CR according to the modified Lugano Criteria for Response Assessment (Cheson 2014)
Time Frame: Up to 18.3 months
Population: The full analysis set includes participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 5 | 6
Percentage of Participants | 20.0 [0.5 to 71.6] | 66.7 [22.3 to 95.7]

8. Secondary Outcome: ORR Per Investigator Assessment According to Modified Lugano Response Criteria
Description: Objective Response Rate (ORR) is defined as the percentage of participants with CR or PR according to the modified Lugano Criteria for Response Assessment (Cheson 2014) based on investigator assessment
Time Frame: Up to 18.3 months
Population: The full analysis set includes participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 5 | 6
Percentage of Participants | 60.0 [14.7 to 94.7] | 83.3 [35.9 to 99.6]

9. Secondary Outcome: DOR Per Investigator Assessment According to Modified Lugano Response Criteria
Description: as for outcome 3
Time Frame: Up to 17.1 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 3 | 5
Months | NA [5.1 to NA] — Not enough events to calculate Median or Upper Limit. | NA [7.2 to NA] — Not enough events to calculate Median or Upper Limit.

10. Secondary Outcome: Progression-free Survival Per Investigator Assessment According to Modified Lugano Response Criteria
Description: as for outcome 5
Time Frame: Up to 18.3 months
Population: The full analysis set includes participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 5 | 6
Months | 6.5 [3.2 to NA] — Not enough events to calculate Upper Limit. | NA [1.1 to NA] — Not enough events to calculate Median or Upper Limit.

11. Secondary Outcome: Rate of Complete Response Per Investigator Assessment According to Modified Lugano Response Criteria
Description: as for outcome 7
Time Frame: Up to 18.3 months
Population: The full analysis set includes participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 5 | 6
Percentage of Participants | 40.0 [5.3 to 85.3] | 66.7 [22.3 to 95.7]

12. Secondary Outcome: ORR Per BICR According to Lugano Response Criteria
Description: ORR is defined as the percentage of participants with CR or PR, assessed according to Lugano Criteria for Response Assessment (Cheson 2014)
Time Frame: Up to 18.3 months
Population: The full analysis set includes participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Classic Hodgkin Lymphoma | PTCL
Number analyzed (Participants) | 5 | 6
Percentage of Participants | 60.0 [14.7 to 94.7] | 83.3 [35.9 to 99.6]

ADVERSE EVENTS:
Time Frame: Non-serious Adverse Events, Serious Adverse Events, and All-Cause Mortality were followed for up to 36 months
Description: The population for All-Cause Mortality includes all enrolled participants. The population for Serious Adverse Events and Other Adverse Events includes participants who received at least one dose of study treatment..
Arm/Group | Classic Hodgkin Lymphoma | PTCL
All-Cause Mortality (participants affected / at risk) | 0/6 | 2/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 2/6
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Classic Hodgkin Lymphoma (N=5) | PTCL (N=6)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Classic Hodgkin Lymphoma (N=5) | PTCL (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3) | 4 (6)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT03947255/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT03947255/SAP_002.pdf